CLINICAL TRIAL: NCT04135222
Title: Evaluation of Periodontal Phenotype Using Cone Beam Computed Tomography (CBCT), Intraoral Scanning by Computed Aided Design (CAD) and Prosthetic-driven Implant Planing (PDIP)
Brief Title: Evaluation of Periodontal Phenotype Using CBCT, Computed Aided Design (CAD) and Prosthetic-driven Implant Planing (PDIP).
Acronym: (CBCT)(CAD)
Status: Completed | Type: Observational
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: kb245/2018
Record Dates: First submitted 2019-09-19; First posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Measurements of gingiva thickness — Measurements were performed at upper canines and incisors in thirty periodontally healthy patients. The CBCT/CAD technology along with the PDIP software were used to measure crestal (CGT in mm ), supracrestal (SGT in mm) and free gingival thickness (FGT in mm ) as well as alveolar crest-gingival margin (AC-GM) and cemento-enamel junction (AC-CEJ) distance and the TLPAC localized 2, 4 and 8mm apically than the edge of the AC. Width of keratinized tissue (WKT) were measured using a periodontal probe. For each patient, the periodontal phenotype was evaluated on the basis of coronal width/length (CW/CL in percentages) ratio of both upper central incisors. For each tooth, the gingival phenotype was assessed on the basis of the GT measurement( in mm).

SUMMARY:
The use of CBCT/CAD and PDIP technology makes it possible to determine the gingival and the periodontal phenotype, and it can be useful in establishing treatment plan in which it is required to carry out radiological diagnostics. Assessment of the periodontal and the gingival phenotype in a patient using the method based on CW/CL ratio is unreliable. Determining it for each dento-gingival unit is the appropriate method.

Positive correlation between FGT, WKT and AC-GM distance confirms the purpose of measuring these parameters for evaluation of the gingival phenotype and additional TLPAC2 for the periodontal phenotype.

DETAILED DESCRIPTION:
The gingival phenotype - (GP) is defined as three-dimensional volume of the gingiva, and is defined by 2 clinical parameters - gingival thickness (GT measured in mm ) and width of keratinized tissue (WKT0measured in mm ). Assessment of the gingival phenotype was performed with the use of visual methods, using the method of gingival transparency while probing the gingival grooves with a periodontal probe, on the basis of transparency of the free gingiva of the upper incisors, the shape of the crowns, the height of gingival papillae, and the width of the gingiva and, recently, using the Colorvue Periodontal Probes. The gingival phenotype may be determined more precisely by using biometry of width of keratinized tissue and gingival thickness. During surgical procedures in which it is planned to form a full thickness flap, GT can be measured in a direct way, for example using an orthodontic caliper or a gauge for thickness of prosthetic crowns measurement. Most often, however, it is advisable to determine the gingival or the periodontal phenotype before initiating dental treatment, at its planning stage.

GT assessment can be performed with the use of invasive methods: with a needle, an endodontic tool or a periodontal probe, with the use of radiological methods - parallel profile radiographs and CBCT, and non-invasive methods - using an ultrasonic device and the optical coherence tomography. Measurements of keratinized tissue width are most often carried out using a periodontal probe calibrated every 1mm.

Assessment of the phenotype is very important not only while planning dental treatment, but also in prediction of its results. A patient with healthy periodontium, but thin phenotype found in a single or in multiple dental units can be protected from the occurrence of complications of orthodontic, prosthetic or implant-prosthetic treatment . Radiological images, obtained by CT scans, are increasingly often assessed while planning such treatment . Scientists have begun to use the possibilities of 3D visualization for the assessment of the periodontal phenotype using the CBCT method.

Assessment of the periodontal and the gingival phenotype in a patient, using the method based on CW/CL, is unreliable. The phenotype should be assessed for each dento-gingival unit.

The presence of positive correlation between WKT, FGT and AC-GM confirms the validity of determining these parameters in the assessment of the gingival phenotype and, additionally, TLPAC2, in determining the periodontal phenotype.

Using the CBCT CAD + PDIP technology allows for determination of the gingival and the periodontal phenotype, and can be useful while planning implantological and orthodontic treatment, in which conducting radiological diagnostics is required. In each case of gingival and periodontal phenotype assessment clinical examination of a patient along with determination of PD, CAL and WKT in the conditions of healthy periodontium should be carried out.

ELIGIBILITY:
Inclusion criteria:

* lack of general diseases
* good hygiene of oral cavity
* healthy periodontium - API ratio<15%, BOP<10%
* no loss of clinical attachment in the examined sites (CAL=0)
* no use of drugs that could influence the structure of the periodontal tissues
* no addictions, especially nicotinism
* no use of mobile prosthetic restorations and orthodontic appliances
* no contraindications for X-ray examinations

Exclusion criteria:

* general diseases
* bad hygiene of oral cavity
* non healthy periodontium - API ratio>15%, BOP>10%
* loss of clinical attachment in the examined sites (CAL>1)
* use of drugs that could influence the structure of the periodontal tissues
* addictions, especially nicotinism
* use of mobile prosthetic restorations and orthodontic appliances
* contraindications for X-ray examinations

Ages: 24 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 16 male 14 female
Study Population: male 16 female 14
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2019-05-13 (Actual); Study Completion 2019-07-07 (Actual)

PRIMARY OUTCOMES:
determination the gingival and the periodontal phenotype | October 2018 to July 2019
  The use of CBCT, CAD and PDIP technology makes it possible to determine the gingival and the periodontal phenotype, and it can be useful in establishing treatment plan in which it is required to carry out radiological diagnostics. Assessment of the periodontal and the gingival phenotype in a patient using the method based on CW/CL (%) ratio is unreliable. Determining it for each dento-gingival unit is the appropriate method.
  Positive correlation between FGT (mm), WKT(mm) and AC-GM (mm) distance confirms the purpose of measuring these parameters for evaluation of the gingival phenotype and additional TLPAC2 for the periodontal phenotype.

CONTACTS AND LOCATIONS:
Overall Officials: wojciech bednarz, prof, Study Director — Medical Uniwersity Wroclaw
Locations (1):
- Wroclaw Medical University, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided